CLINICAL TRIAL: NCT03689790
Title: The Impact of Bariatric Surgery on Estimated Liver Function in Chinese Obesity Patients: a Retrospective Cohort Study
Brief Title: the Related Factors of Bariatric Surgery on Liver Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Jingge Yang, Director of bariatric surgery, First Affiliated Hospital of Jinan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstJinanU20180213
Record Dates: First submitted 2018-06-03; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Liver Function; Bariatric Surgery
MeSH Terms: interventions — Gastric Bypass

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- liver function (Active Comparator): liver function
  Interventions: Procedure: sleeve gastrectomy; Procedure: gastric bypass

INTERVENTIONS:
Procedure: sleeve gastrectomy — sleeve gastrectomy
Procedure: gastric bypass — gastric bypass

SUMMARY:
Obesity and related metabolic diseases have become a chronic disease that is a threat to human health. Bariatric surgery can effectively and long-term reduce excess body weight and relieve related metabolic diseases, including type 2 diabetes. Laparoscopic gastric bypass surgery and laparoscopic sleeve gastrectomy are commonly used in bariatric surgery. Laparoscopic sleeve gastrectomy due to simple operation, good weight loss, and metabolic disease control effect, which is more widely used. However, there are several studies that show an increased chance of gastroesophageal reflux disease after laparoscopic sleeve gastrectomy. Long-term gastroesophageal reflux may lead to Barrett's esophagus or esophageal cancer. Nowadays, the cause of gastroesophageal reflux disease after sleeve gastrectomy is not clear and precautionary measures are not precise.

In this study, prospective randomized controlled trials were conducted to explore the possible causes of liver funnction after bariatric surgery and to explore ways to prevent liver functione after bariatric surgery

DETAILED DESCRIPTION:
With the social development and changes in the lifestyle, the incidence of obesity and type 2diabetes is rapidly increasing. In 2010, the global incidence of type 2 diabetes was 8.3% in adults, 11.6% in China and 50.1% in China. In overweight and obese people, the prevalence of type 2 diabetes also increased significantly, and the prevalence of type 2diabetes in those people with BMI> 30 reached 18.5-23%. Diabetes-induced cardiovascular and cerebrovascular diseases, renal insufficiency and other complications, seriously affecting the quality of life of the patients, endangering the safety of life, the treatment of type 2 diabetes and related complications to public health expenditure has brought tremendous pressure.

Traditional medical methods are difficult to achieve long-term and effective control of type 2 diabetes. Surgery has been shown to achieve 75-95% long-term relief of obesity in patients. Roux-en-Y gastric bypass (Roux-en-Y gastric bypass, RYGB) and laparoscopic sleeve gastrectomy are most commonly used. Among them, laparoscopic sleeve gastrectomy is relatively simple, low incidence of complications, lower operating costs, and gradually become the most important surgical methods of weight loss and metabolic disease surgery. Numerous clinical studies are shown that sleeve gastrectomy in patients with type 2 diabetes has the same therapeutic effect as gastric bypass with a complete remission rate of 70-90% for T2DM.

For the choice of surgical approach, numerous studies have shown that BMI ≧ 45, the general choice of gastric bypass surgery, BMI <45, participants can choose sleeve gastrectomy. The remission rate for T2DM, sleeve gastrectomy has a good result for young patients with shorter duration. In China, the BMI less than 45 is majorities.

According to the previous survey in 2012, the newly diagnosed diabetes patients in China constituted more than half of all diabetic patients. Since bariatric surgery is relatively simple, so bariatric surgery is easier to popularize in China and has wide application prospect.

ELIGIBILITY:
Inclusion Criteria:

* For the choice of surgical approach, numerous studies have shown that BMI ≧ 45, the general choice of gastric bypass surgery, BMI <45, you can choose sleeve gastrectomy. The remission rate for T2DM, sleeve gastrectomy has a good result for young patients with shorter duration. In the investigator's country, the BMI less than 45 is majorities.

Exclusion Criteria:

* BMI<27.5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
preoperative of aminotransferase aspartate | Preoperative
  Aminotransferase aspartate in U/L
Postoperative of aminotransferase aspartate at 3 months | 3 months
  Aminotransferase aspartate in U/L
Postoperative of aminotransferase aspartate at 6 months | 6 months
  Aminotransferase aspartate in U/L
Postoperative of aminotransferase aspartate at 1 year | 1 year
  Aminotransferase aspartate in U/L

SECONDARY OUTCOMES:
preoperative of alanine aminotransferase | Preoperative
  Alanine aminotransferase in U/L
Postoperative of alanine aminotransferase at 3 months | 3 months
  Alanine aminotransferase in U/L
Postoperative of alanine aminotransferase at 6 months | 6 months
  Alanine aminotransferase in U/L
Postoperative of alanine aminotransferase at 1 year | 1 year
  Alanine aminotransferase in U/L

CONTACTS AND LOCATIONS:
Locations (1):
- The frist affiliated hospital of Jinan University, Guangzhou, Guangdong, China